CLINICAL TRIAL: NCT00292357
Title: Local Application of Autologous Bone Marrow Cells for Treatment of Chronic Diabetic Ulcers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD-Med1-01/06
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2007-04

CONDITIONS: Diabetic Foot; Diabetes Complications
MeSH Terms: conditions — Diabetic Foot; Diabetes Complications

INTERVENTIONS:
Procedure: Application of autologous bone marrow

SUMMARY:
Bone marrow cells were previously shown to enhance wound healing in experimental diabetes. In this pilot study, patients with chronic diabetic ulcers not healing under conventional therapy, will be treated with local application of autologous bone marrow cells.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* chronic non-healing foot ulcers (>4weeks)

Exclusion Criteria:

* Charcot foot
* Non-diabetic ulcers
* Ulcers healing under conventional therapy
* Sepsis
* Hematologic disorders
* Pregnancy
* Acute inflammatory disorders
* Chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)

PRIMARY OUTCOMES:
Safety and Feasibility
Healing velocity

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nawroth, MD, Principal Investigator — University of Heidelberg, Dept. Medicine 1, Germany
Locations (1):
- Medizinische Klinik 1, Universitätsklinikum Heidelberg, Heidelberg, Germany